CLINICAL TRIAL: NCT06706856
Title: Quantitative Ultrasound to Assess Steatotic Liver Disease in Children
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Virginia Polytechnic Institute and State University (Other); GE Healthcare (Industry)
Responsible Party: Principal Investigator, Claude Sirlin, Professor of Radiology, University of California, San Diego
Other Study IDs: 809669; 1R01DK135951-01 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: MASLD; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: MASLD; steatosis; quantitative ultrasound; quantitative MRI; fat fraction; PDFF
MeSH Terms: conditions — Fatty Liver | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma, blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort: This is a single arm study in which all participants undergo the same research procedures.
  Interventions: Diagnostic Test: MR exam; Diagnostic Test: US exam; Other: Blood draw; Other: Physical measurements; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: MR exam — Participants will undergo an advanced magnetic resonance (MR) examination of the abdomen and liver.
Diagnostic Test: US exam — Participants will undergo an abdominal ultrasound (US) examination using a full-size US system. Some participants may undergo a point-of-care abdominal US exam with a handheld US system, if possible.
Other: Blood draw — Participants will undergo a blood draw of approximately 25 mL volume.
Other: Physical measurements — Participants will have their height, weight and waist circumference measured. Vital signs including respiratory frequency, heart rate, temperature, and blood pressure will be measured.
Other: Questionnaires — Participants will be asked to fill out questionnaires to collect information about their prescribed medications, demographics, medical and surgical histories, prior laboratory results, physical activity and lifestyle measures, and potential alcohol intake (AUDIT questionnaire).

SUMMARY:
This research study is being conducted to find out more about advanced ultrasound techniques to non-invasively evaluate liver disease in children. The investigators are developing advanced techniques for analyzing ultrasound data and images of the liver, and they will compare it to other established methods used to evaluate the liver, including liver MRI.

The investigators plan to develop and test the advanced analysis techniques using conventional full-size ultrasound machines and, if possible, small handheld devices.

Our goals are:

* To assess the accuracy of the advanced ultrasound analysis techniques in children
* To implement and assess these advanced technique on small handheld ultrasound devices, if possible

DETAILED DESCRIPTION:
Our broad long-term objective is to improve the health of children with metabolic dysfunction-associated steatotic liver disease (MASLD), a condition characterized by accumulation of fat in liver cells, by developing and validating accurate, precise, practical, and widely available tools to detect, measure, and monitor liver fat.

Our study aims to develop advanced quantitative ultrasound (QUS) analysis models for use with full-size US and, if possible, inexpensive point-of-care ultrasound (POCUS) systems in children at risk for MASLD to estimate liver fat fraction and classify presence/absence of fatty liver. We anticipate the models will incorporate technical innovations to improve QUS accuracy and efficiency. To develop and test these models, we plan to enroll 120 children who will undergo ultrasound exams using either full-size or POCUS devices. We plan to compare the performance of our QUS models with liver MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 to 18 years
* Presence of risk factors for having MASLD
* Ability and willingness of participant or legal guardian/parent to give written informed consent
* Participant is willing to give written assent
* Able and willing to undergo all study procedures

Exclusion Criteria:

* Known liver disease other than MASLD
* Pregnant or trying to become pregnant
* Inability to undergo an MR study: weight exceeding scanner table limit, waist circumference > 140 cm, claustrophobie, and/or metal implants.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children being evaluated for MASLD
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Development and Evaluation of models for liver fat estimation. | 5 years
  We plan to develop and evaluate models for estimating liver fat fraction and classifying the presence or absence of steatotic liver disease using QUS data.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Schwimmer, MD, Principal Investigator — University of California, San Diego; Claude B Sirlin, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data and metadata except imaging data will be deposited in the UC San Diego Library Digital Collections Data Repository.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date: 7/1/2025 (anticipated) End date: On or after 7/1/2040 (anticipated)
Access Criteria: The data repository (containing deidentified study data and metadata except imaging data) will be made public and will be available from the UC San Diego Digital Collections Data Repository.
URL: https://library.ucsd.edu/dc